CLINICAL TRIAL: NCT03376087
Title: Cardiac Rhythm Disturbances in Hard-to-treat Epilepsy Patients Using Loop ECG Recorders
Acronym: Epi-Loop-Rec
Status: Completed | Type: Observational
Sponsor: National Research Center for Preventive Medicine (Other Government)
Collaborators: Pirogov Russian National Research Medical University (Other)
Responsible Party: Sponsor
Organization: National Medical Research Center for Therapy and Preventive Medicine (Other Government)
Other Study IDs: 09-04/15 - 6
Record Dates: First submitted 2017-11-28; First posted 2017-12-18 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Epilepsy
Keywords: Epilepsy; heart block; sudden cardiac death; loop recorder
MeSH Terms: conditions — Epilepsy; Heart Block; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Seizure-related cardiac arrhythmias are one of the possible causes of sudden unexpected death in epilepsy (SUDEP). Identification of these patients is challenging because cardiac rhythm disturbances could emerge only during seizures. Furthermore, patients could have transitioned sinus or AV node blocks which could cause syncopes with brady-related seizures which could be treated as epilepsy-related seizures. Implantable loop recorders have an ability to recording single-channel ECG for up to 36 months which give an ability to detect these heart disturbances.

The purpose of this study is to look the incidence and types of arrhythmias which occur in 150 patients with hard-to-treat partial seizures and secondarily generalized seizures

ELIGIBILITY:
Inclusion Criteria:

1. Hard-to-treat focal epilepsy
2. Aged 18 to 60 years
3. If female not pregnant

Exclusion Criteria:

1. Known clinical relevant structural cardiac disease
2. Implanted pacemaker, including cardiac resynchronisation device, or defibrillator
3. Use of beta blockers or other antiarrhythmic medication
4. Diagnosis of psychogenic non-epileptic seizures

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with hard-to-treat epilepsy without known cardiac disease and beta-blockers therapy
Sampling Method: Probability Sample
Enrollment: 193 (Actual)
Dates: Start 2015-11-16 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Identification of a dysrhythmia | 3 years or until the end-of-battery life of Reveal XT, whichever came first
  A dysrhythmia will be defined as either
  * asystole of ≥6 s
  * sinus bradycardia of ≤40 bpm during physical activity
  * 2nd or 3rd-degree AV-block
  * sinus tachycardia of ≥120 bpm
  * nonsustained and sustained monomorphic VT of ≥170 bpm
  * polymorphic VT
  * atrial fibrillation/flutter

SECONDARY OUTCOMES:
The number of patients who will have receive the permanent pacemaker at the end of the study. | 3 years or until the end-of-battery life of Reveal XT, whichever came first

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Serdyuk S, Davtyan K, Burd S, Teryan R, Kharlap M, Drapkina O. A case of sudden unexpected death of a patient with epilepsy: Continuous electrocardiographic monitoring and autopsy results. HeartRhythm Case Rep. 2018 Nov 30;5(3):138-142. doi: 10.1016/j.hrcr.2018.11.014. eCollection 2019 Mar. No abstract available. PMID 30891410
- [Result] Serdyuk S, Davtyan K, Burd S, Drapkina O, Boytsov S, Gusev E, Topchyan A. Cardiac arrhythmias and sudden unexpected death in epilepsy: Results of long-term monitoring. Heart Rhythm. 2021 Feb;18(2):221-228. doi: 10.1016/j.hrthm.2020.09.002. Epub 2020 Sep 8. PMID 32911052